CLINICAL TRIAL: NCT03114332
Title: Subcutaneous Drains In Lean Women Undergoing Cesarean Section, A Randomized Controlled Trial
Brief Title: Subcutaneous Drains And Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Haitham Aboali Hamza, Lecturer of Obstetrics and Gynecology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MU112
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Section

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Patients for whom a subcutaneous drain was used
  Interventions: Procedure: Subcutaneous Drain
- Control group (No Intervention): No drain group

INTERVENTIONS:
Procedure: Subcutaneous Drain — A closed drainage system for the subcutaneous tissue was used (Redivac) through a separate stab wound. Drains were left in place for 24 h or until drainage was less than 50 ml.
  Arms: Study Group

SUMMARY:
A randomized controlled trial that aimed at studying the values (if any) of subcutaneous drains use in lean women during Cesarean section.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most common operative procedures performed in modern obstetrics. Despite being that, common, surgical techniques and steps do widely vary. These variations depend on many factors including surgeons preferences, patient s characteristics and available facilities and circumstances .

The most common complications of Cesarean section are superficial surgical site complications including sepsis, seroma formation and breakdown.

One of the common, yet debatable, practices in Cesarean section is to use a subcutaneous drain for the wound .The advantage of such a practice is to drain any blood or serous fluid that may accumulate in the subcutaneous space, which cause post-operative pain or provide a good medium for microbial growth and infection.

Thus, it is assumed that drains can reduce the burden of surgical site infection. Some surgeons, however, have raised much argument about the value of subcutaneous drains and emerging evidence raised concerns about its effectiveness. Despite this, it is evident that it is still widely used in the clinical practice.

Most randomized controlled trials on this issue, from which we draw the current evidence, were conducted in the developed countries, mainly the United States, with readily available facilities and optimum level of care. This fact raises concerns about how this evidence can be applicable in developing countries with weak health care systems and low level of awareness. In addition, Cesarean section rates are greatly higher in developing countries due to its abuse, which emphasize how the current evidence can't be applicable and in need for further updates .

The current gap between the current practice and lack of evidence has to be filled. In this study, investigators aim at providing answers for this critical issue, thus investigators can ensure women's health and provide the best quality of care following Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. All females with previous cesarean sections admitted to Obstetrics and Gynecology Department at Menoufia University Hospitals either for elective or urgent cesarean section will be considered eligible.

Exclusion Criteria: In order to control any confounding variables, we will exclude women with an added risk of wound complications. Those will include:

1. Diabetic women (as determined by fasting blood sugar and 2-hour Post prandial blood glucose).
2. Morbid obese women (those with body mass index more than 35).
3. Smokers and alcoholics.
4. Immunocompromised women: AIDS patients and those receiving immunosuppressant agents.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of superficial surgical site infection | within 72 hours after the operation
  rate of superficial surgical site infection, defined as presence of wound discharge that yielded a positive result on bacteriological culture within 72 hours after the operation

SECONDARY OUTCOMES:
Wound seroma | up to 6 weeks postoperative
  A seroma is a pocket of clear serous fluid that sometimes develops in the body after surgery
Superficial wound breakdown | up to 6 weeks postoperative
  superficial wound breakdown (defined as skin and/or subcutaneous dehiscence with intact fascial layer)
Postoperative fever | 24 hours postoperatively
  temperature 38 C, 24 hours postoperatively
Postoperative pain | after 24 hours postoperative
  through visual analogue scale (VAS); with 0 meaning no pain, and 10 meaning the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: HAITHAM A HAMZA, MD, Principal Investigator — Menoufia University - Egypt; Ibrahim A Seif El Nasr, MD, Principal Investigator — Menoufia University - Egypt; Nabih I Elkhouly, MD, Principal Investigator — Menoufia University - Egypt
Locations (1):
- Department of Obstetrics and Gynecology - Faculty of Medicine - Menoufia University, Shibīn al Kawm, EL Menofia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Inany H, Youssef G, Abd ElMaguid A, Abdel Hamid M, Naguib A. Value of subcutaneous drainage system in obese females undergoing cesarean section using pfannenstiel incision. Gynecol Obstet Invest. 2002;53(2):75-8. doi: 10.1159/000052996. PMID 11961377
- [Background] Gates S, Anderson ER. Wound drainage for caesarean section. Cochrane Database Syst Rev. 2013 Dec 13;2013(12):CD004549. doi: 10.1002/14651858.CD004549.pub3. PMID 24338262